CLINICAL TRIAL: NCT06171061
Title: Yangxinshi Tablet Intervention for Exercise Capacity in Patients With Chronic Coronary Syndrome: Prospective, Multicentre, Randomized, Open-label, Blinded-endpoint Clinical Trial
Brief Title: Yangxinshi Tablet Intervention for Exercise Capacity in Patients With Chronic Coronary Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong First Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GrowfulPower-008
Record Dates: First submitted 2023-12-05; First posted 2023-12-14 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Chronic Coronary Syndrome
Keywords: Yangxinshi; Chronic Coronary Syndrome
MeSH Terms: interventions — Yangxinshi

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): basic medication + Yangxinshi tablet
  Interventions: Drug: Yangxinshi tablet
- Control group (Other): basic medication.
  Interventions: Other: Basic medication

INTERVENTIONS:
Drug: Yangxinshi tablet — In addition to basic medication, the experimental group will be given Yangxinshi (three tablets each time, three times a day);The treatment period is 24 weeks.
  Other Names: Yangxinshi
  Arms: Experimental group
Other: Basic medication — The control group will be given basic medication only. The treatment period is 24 weeks.
  Arms: Control group

SUMMARY:
This study is a prospective, multicentre, randomized, open-label, blinded-endpoint clinical trial to evaluate the efficacy and safety of Yangxinshi tablets in the treatment of patients with chronic coronary syndrome (CCS).

DETAILED DESCRIPTION:
This study plans to enrol 1200 CCS patients. A central randomized control group will be set up. The experimental and control groups will be populated at a 3:1 ratio. In addition to basic medication, the experimental group will be given Yangxinshi tablets (three tablets each time, three times a day); the control group will be given basic medication only. The treatment period is 24 weeks. The primary efficacy indicator is the 6-minute walking distance (6MWD).

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years;
2. CCS patients in stable condition and clearly diagnosed by coronary artery imaging (at least one vessel stenosis ≥ 50%): stable angina, ischaemic cardiomyopathy, asymptomatic or stable symptoms, occult coronary heart disease, acute coronary syndrome (ACS), or >3 months after coronary revascularization;
3. moderately to severely limited exercise tolerance: the maximum 6MWD is < 450 m, or the metabolic equivalent (MET) as measured by treadmill cardiopulmonary exercise testing is < 5 METs;
4. voluntary participation and signing of informed consent.

Exclusion Criteria:

1. absolute or relative contraindications for the treadmill cardiopulmonary exercise test or 6-minute walk test (6MWT);
2. serious primary diseases, mental diseases, or malignant tumours that affect lifespan;
3. pregnancy, intended or suspected pregnancy, miscarriage, breastfeeding, or delivery in the last 6 months;
4. subjects not suitable for this study in the opinion of the researchers, such as subjects who are participating in other drug clinical trials or intervention studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
6MWD | 24 weeks after treatment
  The 6-min walking distance

SECONDARY OUTCOMES:
Borg scale | 24 weeks after treatment
  score range: 0~10,higher scores mean a worse outcome.
MACCE | after 4, 8, 12, 16, 20, and 24 weeks of treatment
  incidence of major adverse cardiovascular and cerebrovascular events (MACCE)

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Haitao, Principal Investigator — Shandong Provincial Hospital
Locations (32):
- China (32):
  - Shapingba District People's Hospital of Chongqing, Chongqing, Chongqing Municipality
  - Zhengzhou Seventh People's Hospital, Zhengzhou, Henan
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Binzhou People's Hospital, Binzhou, Shandong
  - Dezhou Municiple Hospital, Dezhou, Shandong
  - Pingyuan County first People's Hospital, Dezhou, Shandong
  - Feicheng People's Hospital, Feicheng, Shandong
  - Shandong Health Group Feicheng Hospital, Feicheng, Shandong
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Jinan Zhangqiu District People's Hospital, Jinan, Shandong
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - The Fourth People's Hospital of Jinan, Jinan, Shandong
  - Gaotang County People's Hospital, Liaocheng, Shandong
  - Liaocheng Hospital of Traditional Chinese Medicine, Liaocheng, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - The Second People's Hospital of Liaocheng, Liaocheng, Shandong
  - Linqing City People's Hospital, Linqing, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Longkou People Hosptial, Longkou, Shandong
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Hospital of Cardiovascular Diseases Affiliated to Qingdao University, Qingdao, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Qingdao Fuwai Hospital, Qingdao, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Shandong University Qilu Hospital Qingdao District, Qingdao, Shandong
  - The Second Affiliated Hospital of Shandong First Medical University, Taian, Shandong
  - Xintai People's Hospital, Taian, Shandong
  - Tengzhou Central People's Hospital, Tengzhou, Shandong
  - Weifang City People's Hospital, Weifang, Shandong
  - Weifang City Yidu Central Hospital, Weifang, Shandong
  - Yantai Hospital of Traditional Chinese Medicine, Yantai, Shandong